CLINICAL TRIAL: NCT04981522
Title: Indigenously Adapted Community Based Psychological Intervention for Individuals Living with Disabilities: a Cluster Randomized Clinical Trial
Brief Title: Community Based Psychological Intervention for Persons Living with Disabilities
Acronym: CBPI-PWD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Islamic University, Islamabad (Other)
Collaborators: Aid To Leprosy Patients (ALP), Rawalpindi-Pakistan (Unknown)
Responsible Party: Principal Investigator, Basharat Hussain, Lecturer/PhD Scholar, International Islamic University, Islamabad
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 64-FSS/PHDPSY/F18
Record Dates: First submitted 2021-07-19; First posted 2021-07-29 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-03

CONDITIONS: Physical Condition, Minor Psychological Component; Psychological Distress

STUDY DESIGN:
Intervention Model Description: Research design of the study shall consists of two-arms, single-blind cluster randomized controlled trial (c-RCT). While Randomized Control Trial (RCT) shall consists of two groups: Active Treatment (AT) and Delayed Treatment Control (DTC).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Single-blind cluster randomized controlled trial (c-RCT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Treatment (AT): PM+ intervention (Experimental): Active Treatment (AT) group will receive 05 sessions of indigenously adapted problem management plus (IA-PM+) intervention.
  Interventions: Behavioral: Indigenously adapted problem management plus (IA-PM+)
- Delayed Treatment Control (DTC): Treatment as usual (No Intervention): Delayed Treatment Control (DTC) group will receive routine treatment until the last follow-up.

INTERVENTIONS:
Behavioral: Indigenously adapted problem management plus (IA-PM+) — The IA-PM+ manual would be comprised of the following evidence-based techniques: (a) problem solving, (b) stress management, (c) behavioral activation and (d) accessing social support. The IA-PM+ intervention consisting of five sessions, will teach the participants techniques to manage their emotional problems.
  Other Names: Problem management plus (PM+)
  Arms: Active Treatment (AT): PM+ intervention

SUMMARY:
Mental health problems are increasing in Pakistan and there is a 90% treatment gap in mental health services. Accessibility towards mental health services is limited due to range of factors including low income and resources, lack of the trained staff and lack of specialized and non-specialized mental health facilities. Therefore, there is a dire need to develop indigenous solution of the mental health issues grounded in Islamic teaching.

In this regard this study is designed to address the mental health issues at community level. Therefore, this study divided into two phases. In first phase the aim of the study is to adapt World Health Organization recommended psychological intervention for paraprofessionals and to train the paraprofessional on this indigenously adapted intervention. Subsequently, in second phase the study aims to assess the effectiveness of the indigenously adapted Problem Management Plus (IA-PM+) as an evidence based remedy in the treatment of psychological distress of person living with disabilities (PWDs).

DETAILED DESCRIPTION:
Prevalence of disability is higher in Low and middle income countries (LMICs). Persons living with disabilities are more vulnerable to develop psychopathology due to their low level of functioning, their complex and speciﬁc needs. Consequently, Persons living with disabilities (PWDs) are expected to experience more adverse psychological ailments as compared to the persons living without disabilities particularly in the rural parts of the countries. Accessibility towards mental health services in Pakistan has been limited due to range of factors including low income and resources, lack of the trained staff and lack of specialized and non-specialized mental health facilities. These challenges are required to be dealt at locally at micro and macro levels systemically and effectively. This requires development and innovation in the existing infrastructure by devising multidisciplinary community based treatment policy in building mental health care services. Therefore, to integrate the mental health care services at primary care level, there is a dire need to develop indigenous psychological interventions in a simplified form so that people can quickly learn their utilization not only from the health professionals but also from the para-professionals as well.

Due to the lack of specialized mental health services and human resources in low resource settings, task shifting is a well-known strategy, designed by World Health Organization to bridge the treatment gap in mental health problems. This strategy empowers the health workers, such as nurses and non-specialist to perform specific roles to bridge the available treatment gap. In addition to this, deliverance of evidence based psychological treatment by para-professionals/ non-specialists will not only help in reducing the financial and human resources but also might be able to reduce the stigma associated with mental illness.

Realizing the influence of religion on the general population, the American Psychological Association (APA) has recommended to view the religion as a significant aspect of human life and as such psychologists need to get special knowledge and training on religious psychotherapy.

In this regard this study is designed to address the mental health issues at community level. Therefore, this study divided into two phases. In first phase the aim of the study is to adapt World Health Organization recommended psychological intervention for paraprofessionals and to train the paraprofessional on this indigenously adapted intervention. Subsequently, in second phase the study aims to assess the effectiveness of the indigenously adapted Problem Management Plus (IA-PM+) as an evidence based remedy in the treatment of psychological distress of person living with disabilities (PWDs).

ELIGIBILITY:
Inclusion Criteria:

* Score more than 16 (16>) On PSYCHLOPS
* Participants living with permanent disabilities (more than 6 months)

Exclusion Criteria:

* Temporary resident or people living outside the study area.
* Participants who are unable to engage or respond to the research question
* Diagnosed psychiatric patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
WHO Disability Assessment Scale (WHODAS 2.0) | Assessments will be conducted at baseline (after the screening), 8th week (2 month) after the baseline, 20th week (5th month) after the baseline. The purpose of the outcome measure is to asses the change from baseline to follow-up.
  WHODAS 2.0 is a self-report instrument is used to assess health and disability. The WHODAS assess people's difficulties associated to their illness across six domains of functioning (mobility, cognition, self-care, getting along, life activities and participation). Its five-point Likert scale keeps record of the last 30 days. The 12-item WHODAS 2.0 version translated in Urdu will be used in this study. (World-Health-Organization, 2010).
Depression Anxiety Stress Scale (DASS-21) | Assessments will be conducted at baseline (after the screening), 8th week (2 month) after the baseline, 20th week (5th month) after the baseline. The purpose of the outcome measure is to asses the change from baseline to follow-up.
  DASS is a 21 items Likert-scale is used to assess the possibility of depression, anxiety and stress among the study population (Lovibond & Lovibond, 1995).

SECONDARY OUTCOMES:
Multidimensional Scale of Perceived Social Support (MSPSS) | Assessments will be conducted at baseline (after the screening), 8th week (2 month) after the baseline, 20th week (5th month) after the baseline.
  MSPSS measures perceived social support. Its seven point Likert scale, includes 12 items that cover three dimensions: family, friends and other significant.
Satisfaction with Life Scale (SWLC) | Assessments will be conducted at baseline (after the screening), 8th week (2 month) after the baseline, 20th week (5th month) after the baseline.
  Satisfaction with Life Scale (SWLC) is a 5-item scale designed to measure the global cognitive judgements of one's life satisfaction.
Client Satisfaction Questionnaire (CSQ) | The questionnaire will be employed on the 8th week (2 month) after the baseline and at the 20th week (5th month) after the baseline.
  The Client Satisfaction Questionnaire is a brief and simple scale to measure the patient satisfaction with mental health services.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Muhammad Tahir Khalily, PhD, Study Chair — International Islamic University, Islamabad
Locations (1):
- Community Based Inclusive Development (CBID) Center, Basic Health Unit (BHU) Kuri Dolal, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamdani SU, Ahmed Z, Sijbrandij M, Nazir H, Masood A, Akhtar P, Amin H, Bryant RA, Dawson K, van Ommeren M, Rahman A, Minhas FA. Problem Management Plus (PM+) in the management of common mental disorders in a specialized mental healthcare facility in Pakistan; study protocol for a randomized controlled trial. Int J Ment Health Syst. 2017 Jun 8;11:40. doi: 10.1186/s13033-017-0147-1. eCollection 2017. PMID 28603552
- [Background] Some D, Edwards JK, Reid T, Van den Bergh R, Kosgei RJ, Wilkinson E, Baruani B, Kizito W, Khabala K, Shah S, Kibachio J, Musembi P. Task Shifting the Management of Non-Communicable Diseases to Nurses in Kibera, Kenya: Does It Work? PLoS One. 2016 Jan 26;11(1):e0145634. doi: 10.1371/journal.pone.0145634. eCollection 2016. PMID 26812079
- [Background] Iemmi, V., Gibson, L., Blanchet, K., Kumar, K. S., Rath, S., Hartley, S., . . .Kuper, H. (2014). Community-based rehabilitation for people with disabilities in low-and middle-income countries: A systematic review. Campbell Systematic Reviews, 11(1), 1-177.
- [Background] Hussain B, Khalily MT, Hallahan B. Psychological intervention for a person living with amblyopia: a case study from home-based integrated care. J Pak Med Assoc. 2023 Jun;73(6):1330-1333. doi: 10.47391/JPMA.7304. PMID 37427645
- [Background] Hussain, B., & Khalily, M. T. (2024). Enhancing Community Resilience: integrated home-based psychological intervention for individuals living with physical disabilities. Journal of Professional & Applied Psychology, 5(1)
- [Background] Hussain, B., Khalily, M. T., & Zaman, S. (2024). Integrated Psychological Intervention for Amelioration of Mental Health Problems of Individuals with Physical Disabilities in Pakistan. Al-Qirtas, 3(1), 159-167.
- [Derived] Hussain B, Khalily MT, Waqas A, Rahman A, Angelakis I, Nisar A, Zaman S, Akhtar T. Acceptability and efficacy of the culturally adapted problem management plus intervention for people with disability in Pakistan: a pilot cluster randomized controlled trial. Front Psychiatry. 2025 Jan 30;15:1413809. doi: 10.3389/fpsyt.2024.1413809. eCollection 2024. PMID 39980593
- See also: Related Info — https://www.frontiersin.org/journals/psychiatry/articles/10.3389/fpsyt.2024.1413809/abstract